CLINICAL TRIAL: NCT00829192
Title: A Multicentre, Randomised, Double-Blind, Placebo Controlled, Phase II Study to Evaluate the Safety and Efficacy of Subcutaneous Bioresorbable Implants of Afamelanotide (CUV1647) for the Prophylactic Treatment of Pre-Cancerous Skin Lesions of the Head, Forearms and Hands in Immune Compromised, Organ Transplant Patients.
Brief Title: Phase II AK Study in Organ Transplant Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Clinuvel Pharmaceuticals Limited (Industry)
Responsible Party: Dr Dennis Wright, Clinuvel Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CUV011
Record Dates: First submitted 2009-01-23; First posted 2009-01-26 (Estimated); Last update posted 2010-12-06 (Estimated); Status verified 2010-12

CONDITIONS: Actinic Keratoses; Carcinoma, Squamous Cell; Organ Transplant Recipients
Keywords: Actinic keratoses (AK); Squamous cell carcinomas (SCC); CUV1647; Afamelanotide; Clinuvel; Photoprotection; Organ transplant
MeSH Terms: conditions — Keratosis, Actinic; Carcinoma, Squamous Cell | interventions — afamelanotide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Afamelanotide (CUV1647) implant administered subcutaneously every 60 days for 24 months
  Interventions: Drug: Afamelanotide (CUV1647)
- 2 (Placebo Comparator): Placebo implant administered subcutaneously every 60 days for 24 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Afamelanotide (CUV1647) — 16 mg subcutaneous implant administered every 60 days
  Arms: 1
Drug: Placebo — Placebo subcutaneous implant administered every 60 days
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether afamelanotide (CUV1647) is effective in reducing the number of actinic keratoses and squamous cell carcinomas developing in immune compromised organ transplant recipients, who are at particularly high risk, over a 24 month test period.

The number of lesions formed on the head, hands and forarms will be monitored over this 24 month test period.

ELIGIBILITY:
Inclusion Criteria:

* Organ transplant recipients with stable transplant function and who received their transplant at least 2 years prior to study entry
* Organ transplant patients who have had at least one biopsy-positive SCC
* Aged 18 - 75 years
* Written informed consent to the performance of all study-specific procedures

Exclusion Criteria:

* Allergy to afamelanotide (CUV1647) or the polymer contained in the implant
* History of melanoma
* Current pigmentary disorders such as melasma
* Diagnosed with HIV/AIDS, or hepatitis B or C
* Current history of drug or alcohol abuse (in the last 12 months)
* Clinically significant organ dysfunction, history of medical disorders or other factors, which in the opinion of the investigator will interfere with the interpretation of study outcome measures
* Major medical or psychiatric illness
* Pregnancy as confirmed by positive serum beta-HCG pregnancy test prior to baseline or lactating mothers
* Females of child bearing potential not using adequate contraceptive measures
* Participation in a clinical trial for an investigational agent within 30 days prior to the screening visit
* Use of regular medications or any other factors that may affect skin pigmentation

Discontinuation Criteria:

* Initiation of treatment with systemic retinoids
* Change of class of systemic immunosuppressant treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2007-11; Primary Completion 2012-07 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
To determine the effect of afamelanotide (CUV1647) administered from slow release subcutaneous implants on the number of actinic keratoses (AKs) on the head, forearms and back of hands | 24 months

SECONDARY OUTCOMES:
To determine and compare the proportion of patients in each group that develops one or more squamous cell carcinoma (SCC) | 24 months
To examine the effect of ongoing sun exposure on lesion formation and progression in the patient group | 24 months
To evaluate the safety and tolerability of multiple slow release subcutaneous implants of afamelanotide (CUV1647) | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Günther Hofbauer, M.D., Principal Investigator — Universitätsspital Zürich
Locations (12):
- Australia (3):
  - The Princess Alexandra Hospital, Brisbane, Queensland
  - The Queen Elizabeth Hospital, Adelaide, South Australia
  - The Royal Melbourne Hospital, Melbourne, Victoria
- Belgium (2):
  - Hospital Erasme, Brussels
  - Gent University Hospital, Ghent
- University Hospital, Besançon, France
- Germany (2):
  - Charité Univeritätsklinikum, Berlin
  - Kiel University Hospital, Kiel
- Italy (2):
  - Ospedali Riuniti di Bergamo, Bergamo
  - University of Padua, Padua
- Karolinska University Hospital, Stockholm, Sweden
- Universitätsspital Zürich, Zurich, Switzerland